CLINICAL TRIAL: NCT03767803
Title: Collection of Whole Blood Samples for the Evaluation of Preeclampsia (Pre-E) Biomarkers
Brief Title: Collection of Whole Blood Samples for the Evaluation of Preeclampsia (Pre-E) Biomarkers From Pregnant Women
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Progenity, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO-129-PREECLAMPSIA
Record Dates: First submitted 2018-12-05; First posted 2018-12-07 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Pre-Eclampsia; Hypertension; Proteinuria in Pregnancy; Thrombocytopenia; Renal Insufficiency; Impaired Liver Function; Pulmonary Edema; Headache; Visual Impairment
Keywords: Hypertension; Proteinuria; Thrombocytopenia; Renal Insufficiency; Impaired Liver Function; Pulmonary Edema; Cerebral Symptoms; Visual Symptoms
MeSH Terms: conditions — Pre-Eclampsia; Hypertension; Thrombocytopenia; Renal Insufficiency; Liver Diseases; Pulmonary Edema; Headache; Vision Disorders; Proteinuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — This study will collect 20 mL whole blood samples from subjects at one or more study visits. The whole blood will be processed to plasma and stored for testing.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Positive Preeclampsia group: A group with diagnosis of preeclampsia within 24 hours of testing and pre-term delivery
  Interventions: Other: Non-interventional study
- Study Cohort: A group without diagnosis of preeclampsia. Also includes a group without diagnosis of preeclampsia within 24 hours of testing, but who have subsequent worsening or re-emergence of signs and symptoms of preeclampsia, and are later diagnosed with preeclampsia and have pre-term delivery.
  Interventions: Other: Non-interventional study

INTERVENTIONS:
Other: Non-interventional study — This is an observational, non-interventional study.

SUMMARY:
Whole blood sample procurement study from pregnant women with signs and symptoms of Preeclampsia.

DETAILED DESCRIPTION:
This multicenter non-interventional observational sample acquisition study is designed to acquire whole-blood samples from pregnant women who present with signs and symptoms of Pre-E and are in the care at an OB-GYN and/or Maternal Fetal Medicine (MFM) site, defined as outpatient centers, clinic sites, and medical offices.

Study population includes subjects who are pregnant, of any race or ethnicity, 18 to 45 years of age, 28 0/7 to 36 6/7 weeks' gestational age with a singleton fetus and have provided written informed consent to provide whole blood specimens at one or more study visits.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 to 45 years of age
* Subject is willing to provide informed consent
* Subject enrolling at a study OB-GYN or MFM site is in the opinion of the physician able to provide 20 mL of whole blood and will comply with all study procedures
* Subject has a singleton fetus of 28 0/7 to 36 6/7 weeks' gestational age using 2014 ACOG Dating Criteria (pregnancies starting as twins but complicated with either vanishing twin syndrome or fetal demise of one twin before 14 weeks, are eligible for inclusion)
* Patient presenting with clinical suspicion of Pre-E based on one or more of the following clinical signs and symptoms of Pre-E:

  * New onset increased blood pressure in otherwise normotensive patient
  * Worsening hypertension in a patient with pre-existing hypertension
  * New onset proteinuria or worsening of pre-existing proteinuria
  * Any other clinical finding typically associated with suspicion of Pre-E and requiring workup to rule-out Pre-E

Exclusion Criteria:

* Pregnancy is non-viable, as evidenced by absence of fetal cardiac activity
* Major fetal anomaly or chromosomal aneuploidy
* Current dialysis for kidney failure, including continuous ambulatory peritoneal dialysis

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Subjects who are pregnant, of any race or ethnicity, 18 to 45 years of age, 28 0/7 to 36 6/7 weeks' gestational age with a singleton fetus and have provided written informed consent to provide whole blood specimens at one or more study visits.
Sampling Method: Non-Probability Sample
Enrollment: 344 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of preeclampsia is determined by standard of care. | 3 months
  Observational, non-interventional sample procurement study in which participants are treated per standard of care

CONTACTS AND LOCATIONS:
Overall Officials: Peter Stiegler, PhD, Study Director — Progenity, Inc.
Locations (24):
- United States (24):
  - West Coast Medical Research, Inc., San Diego, California
  - Christiana Care, Newark, Delaware
  - Women's Health Partners, LLC, Boca Raton, Florida
  - Discovery Clinical Research, Plantation, Florida
  - Leavitt Clinical Research, Idaho Falls, Idaho
  - Norton Healthcare, Louisville, Kentucky
  - Obstetrics and Gynecology Associates AMB, Silver Spring, Maryland
  - Valley OB-GYN Clinic, PC, Saginaw, Michigan
  - Rutgers-RWJMS, New Brunswick, New Jersey
  - St. Peter's University Hospital, New Brunswick, New Jersey
  - Virtua Voorhees Hospital, Voorhees Township, New Jersey
  - New Life Medical Esthetics and Wellness, PLLC, Brooklyn, New York
  - Columbia University, New York, New York
  - Total Woman Care, Elkin, North Carolina
  - David B. Schwartz, MD, LLC, Cincinnati, Ohio
  - Obstetrics & Gynecology Associates, Inc., Fairfield, Ohio
  - Hilltop Obstetrics & Gynecology, Franklin, Ohio
  - Dr. Ahuja and Associates OB-GYN, Mentor, Ohio
  - Drexel University, Philadelphia, Pennsylvania
  - The Jackson Clinic, PA, Jackson, Tennessee
  - Aa Ob-Gyn, Pllc, Austin, Texas
  - OB-GYN North, Austin, Texas
  - Corpus Christi Women's Clinic, Corpus Christi, Texas
  - Advanced Clinical Research, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No